CLINICAL TRIAL: NCT05316467
Title: Weight Management Plus Megestrol Acetate in Early-stage Endometrioid Carcinoma: Two Single-arm, Prospective and Open-label Clinical Study
Brief Title: Weight Management Plus Megestrol Acetate in Early-stage Endometrioid Carcinoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, MD.PhD. Vice president of Obstetrics & Gynecology Hospital of Fudan University, Fudan University
Organization: Fudan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53211036-01
Record Dates: First submitted 2022-03-09; First posted 2022-04-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Carcinoma; Obese; Overweight; Fertility Issues
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Overweight; Infertility | interventions — Megestrol Acetate; Tablets

STUDY DESIGN:
Intervention Model Description: All enrolled patients will receive enhanced lifestyle management to control weight and take Megestrol Acetate (MA) for treating EEC.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- overweight 24kg/m2≤BMI<28kg/m2 (Experimental): MA+ weight management enrolled patients will receive megestrol acetate 160mg po qd plus weight management
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI); Drug: Megestrol Acetate 160 MG Oral Tablet
- BMI≥28kg/m2 (Experimental): MA+ weight management enrolled patients will receive megestrol acetate 160mg po qd plus weight management
  Interventions: Behavioral: Intensive Lifestyle Intervention (ILI); Drug: Megestrol Acetate 160 MG Oral Tablet

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention (ILI) — * dietary guidance
  * exercise guidance
  * lifestyle intervention
  Other Names: Weight Management
Drug: Megestrol Acetate 160 MG Oral Tablet — enrolled participants will take Megestrol Acetate 160mg daily
  Other Names: yilizhi

SUMMARY:
To investigate the efficacy of weight management plus megestrol acetate in obese patients with early endometrioid carcinoma（EEC）asking for fertility-sparing treatment

DETAILED DESCRIPTION:
Background:

High-dosage high-efficacy progesterone, such as Megestrol Acetate (MA) and medroxyprogesterone acetate(MPA), is still the first-line treatment for women with early endometrioid endometrial cancer (EEC) who want to preserve fertility. Approximately 70% to 80% of females who meet the criteria for conservation treatment are able to achieve CR after progestin therapy, with a median time of 6-7 months, but about 20% to 30% of patients get no response or need to take longer time to achieve remission (over one year). Overweight/obesity is an independent risk factor for fertility-sparing treatment response and pregnant outcomes in young females with early endometrioid cancer, substantial evidence showed that obesity can cause relatively lower complete response（CR）rates, longer time to achieve completer remission and lower birth rates besides metabolic disorders and other adverse effects caused by obesity. Weight management has been found to improve metabolic disorders, ovarian functions and pregnant outcomes.The hypothesize is that weight management plus progestin therapy may raise CR rates and pregnant outcomes in young female EEC patients asking for fertility conservation. Previous research has shown that metformin plus MA can increase CR rates. Enhanced lifestyle management (diet control, exercise and daily behavioral guidance) may improve metabolic conditions, increase CR rates and pregnant outcomes in obese EEC patients who want to preserve fertility. Till now, no similar studies were found, so the investigators design this study to explore the efficacy of weight control in EEC fertility-sparing patients to provide new evidence for improving conservative treatment.

Objective: To investigate whether weight management plus MA improve the efficacy of preserving fertility when compared to MA alone in obese women with EEC who want fertility conservation.

Design: This study is two single-arm, prospective, open-label. Patients with early-stage endometrioid carcinoma requiring conservation treatment with BMI ≥ 24 kg/m2 will be recruited in this study and they will be divided into two arms, one is overweight group (24kg/m2≤BMI<28kg/m2) and another is obese group (BMI≥28kg/m2). Each arm and its sample size was designed according to Simon's Two-Stage Design. All enrolled patients will receive enhanced lifestyle management to control weight and take MA for treating EEC. Hysteroscopic examination, metabolic and inflammatory indicators will be performed every 12 to16 weeks while other indexes will be evaluated every month, including weight, heart rates，blood pressure and so on.For the progestin efficacy evaluation, CR is defined as the remission of EEC to proliferative or secretory endometrium; partial response (PR) is defined as regression to simple or complex hyperplasia with or without atypia; no response (NR) is defined as the persistence of the disease; and progressive disease (PD) is defined as disease progression in patients. Two months' maintenance treatment will be recommended for patients with CR, and participants will be followed up for 2 years.

Outcomes: Primary outcome is the CR rates of the two arms (overweight and obesity group). Secondary outcomes include pregnancy rates, live birth rates, weight loss, insulin resistance, chronic inflammation indicators, time to achieve CR and the recurrence rates and so on. Safety and side events during the whole trial will be monitored in two years.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years≤age≤45years
2. BMI (body mass index) ≥24kg/m2
3. Consent informed and signed
4. Pathologically confirmed as endometrial carcinoma Patients with endometrial specimens obtained by endometrial biopsy, diagnostic curettage or hysteroscopy and diagnosed histologically as endometrioid carcinoma, G1. If specimens are from other hospitals, they must be counseled or reconfirmed by the Department of Pathology of the Obstetrics and Gynecology Hospital of Fudan University.
5. Imaging Assessment Enhanced MRI of the pelvis and enhanced CT of the upper abdomen must be performed in 2 weeks prior to starting treatment to assess the lesions confined to the endometrial layer without clear myometrial infiltration or extrauterine involvement.
6. Have a strong desire to reproduce and ask for fertility preservation or those who insist on keeping the uterus despite no reproductive requirements.
7. Have good compliance and follow-up conditions, and patients are willing to follow up in Obstetrics and Gynecology Hospital of Fudan University in time.

Exclusion Criteria:

1. Patients with non-endometrioid endometrial carcinoma, endometrioid endometrial carcinoma G2/G3 or other malignant tumors of the reproductive system; imaging suggests myometrial invasion, cervical involvement or extra-uterine involvement.
2. Combined with severe medical disease or liver or kidney dysfunction: alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels elevate to 3 times or more of the upper limit of normal, kidney dysfunction (creatinine clearance <30 mL/min)
3. Patients with other types of endometrial cancer or other malignant tumors of the reproductive system; patients with breast cancer or other hormone-dependent tumors that cannot be used with progesterone.
4. Those who have received high doses of high potency progestin or oral contraceptives within the last 3 months (or those on maintenance medication).
5. Those who require hysterectomy or other methods other than conservative treatment.
6. Known or suspected pregnancy.
7. Those who has contraindications to use progestin.
8. Deep vein thrombosis, stroke, myocardial infarction.
9. Severe joint lesions that prevent walking or movement.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (CR) rates | From date of recruitment until the date of CR, assessed up to 28 weeks.
  The 28-week CR rates will be calculated in two arms

SECONDARY OUTCOMES:
Pregnancy outcomes | up to 2 years after complete response of the last participant
  For patients have a desire for fertility, pregnancies, births and related outcomes will be counted, and the rate of pregnancy will be counted as number of pregnancies/ number of patients trying to fertility in the following period.
Weight change | From date of recruitment, assessed up to 28 weeks.
  Body weight will be recorded every month and compare its change during the trial in kilograms.
Change of body composition | From date of recruitment, assessed up to 28 weeks.
  Assess the improvement of body composition, the investigators will detect body composition with InBody machine and calculate changes of the indicated indexes.
Change of heart rates | From date of recruitment, assessed up to 28 weeks.
  Record heart rates in bpm (beats per minute) every 12-16 weeks and calculate its change during the trial.
Change of blood pressures | From date of recruitment, assessed up to 28 weeks.
  Record blood pressure (both of systolic and diastolic pressures) every 12-16 weeks and compare its change during the treatment.
Blood glucose change | From date of recruitment, assessed up to 28 weeks.
  Assess fasting glucose levels each 3 to 4 months and calculate changes during the trial in mmol/L.
Blood lipids change | From date of recruitment, assessed up to 28 weeks.
  Assess blood lipids levels each 3 to 4 months and compare their change during the treatment.
Insulin resistance change | From date of recruitment, assessed up to 28 weeks.
  Assess fasting insulin levels each 3 to 4 months and compare their changes during the trial.
Ovarian reserve function change | From date of recruitment, assessed up to 28 weeks.
  Detect serum Anti-Mullerian Hormone (AMH) levels each 3 or 4 months and calculate its change.
Quality of life change | From date of recruitment, assessed up to 28 weeks.
  Collect quality of life questionnaire (SF-36 and IWQOL-LITE) every 12-16 weeks and count scores.
Physical activities change | From date of recruitment, assessed up to 28 weeks.
  Collect physical activities questionnaire（IPAQ）and compare scores changes through conservative treatment.
Chronic inflammatory indexes change | From date of recruitment, assessed up to 28 weeks.
  Detect chronic inflammatory indexes, including TNF-α(tumor necrosis factor), IL-1 and IL-6, and calculate changes through the whole treatment period.
Time of pathological complete response (CR) | From date of recruitment until the date of CR, assessed up to 2 years.
  Time of histologic regression from EC to proliferative or secretory endometrium
Incidence of adverse events | From date of recruitment until the date of CR, assessed up to 2 years.
  Adverse events related with MA and weight control. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Relapse rates | up to 2 years after the treatment for each patient
  All enrolled patients will be followed up for 2 years. During the following-up period, if patients recur after complete regression, they will be counted and the number of recurrence will be divided by number of patients followed up, then the investigators can get the relapse rates. Comparison will be performed between two groups.

CONTACTS AND LOCATIONS:
Overall Officials: XIAOJUN CHEN, PhD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No